CLINICAL TRIAL: NCT06680453
Title: Accidentology and Traumatology Associated With Foiling in Brittany
Acronym: TRAUMAF
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Brest (Other)
Collaborators: Centre Hospitalier des Pays de Morlaix (Other); Hospital, Quimper (Unknown); Centre Hospitalier de Bretagne Sud (Other); Hospital, Douarnenez (Unknown)
Responsible Party: Sponsor
Other Study IDs: 29BRC24.0152
Record Dates: First submitted 2024-10-16; First posted 2024-11-08 (Actual); Last update posted 2025-01-22 (Actual); Status verified 2024-11

CONDITIONS: Sport Injuries

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
In the 2010s, the practice of water sports was turned upside down by the arrival of a new discipline: foiling. The number of sailors, particularly amateurs, is increasing every every year. The foil offers greater speed and height, and has therefore the accidents and injuries that result. injuries. But there are very few studies on the subject. The TRAUMAF study proposes to compare the distribution of the number of patients injured during water sports with and without the use of foils. The study also looks at patient management and the type of injury. The aim is to anticipate the management of these patients during periods of practice of these sports.

Translated with DeepL.com (free version)

ELIGIBILITY:
Inclusion Criteria:

* Patient of legal age
* Patient not expressing refusal to participate in the study
* Patient consulting an emergency room following a boating accident that occurred no more than 7 days previously
* Patient able to complete a questionnaire

Exclusion Criteria:

* Minor patient
* Patients who are illiterate and/or do not understand French
* Patient under legal protection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Any person of legal age, meeting the inclusion and non-inclusion criteria, presenting to an emergency department following a boating accident.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2025-01-15 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Evaluate the importance of foil-equipped craft in the occurrence of water-related injuries. | 12 months
  Percentage of boating accidents involving foils.

SECONDARY OUTCOMES:
Provide the doctor in charge of the patient with objective data on the most likely lesions and their potential severity. | 12 months
  Distribution of the frequency of different types of injury according to whether or not the foil was used (comparison between the two study groups).
Analysis of the type and location of lesions observed between the foil and no-foil groups. | 12 months
  Comparison of the location of injuries observed between the foil and non-foil groups. Comparison of accident type (fall, cut, impact, etc.) between the two groups.

CONTACTS AND LOCATIONS:
Locations (5):
- France (5):
  - CHU de Brest, Brest, Finistère
  - Centre Hospitalier Michel Mazéas, Douarnenez, Finistère
  - Centre Hospitalier de Morlaix, Morlaix, Finistère
  - Centre Hospitalier Intercommunal de Cornouaille, Quimper, Finistère
  - GHBS Hôpital du Scorff, Lorient, Morbihan